CLINICAL TRIAL: NCT05501340
Title: Phase I-II Clinical Study of PRaG（PD-1 Inhibitor Intravenous Injectio,Radiotherapy and GM-CSF）Combined With PD-1 Inhibitor Intraperitoneal Perfusion for Advanced Refractory Solid Tumors Combined With Malignant Ascites
Brief Title: PD-1 Inhibitor Intraperitoneal Perfusion Combined With PRaG Therapy for Malignant Ascites
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2022-033-02
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Malignant Ascites
MeSH Terms: interventions — molgramostim; regramostim

STUDY DESIGN:
Intervention Model Description: Intraperitoneal infusion of PD-1 inhibitor can produce anti-tumor effect, and intraperitoneal infusion of PD-1 inhibitor combined with PRaG（Radiotherapy and GM-CSF）can benefit the survival of patients with peritoneal metastasis of advanced malignant tumors and malignant ascites
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRaG combined PD-1 inhibitor intraperitoneal injection (Experimental): PRaG(PD-1 inhibitor,Radiotherapy and GM-CSF) combined with PD-1 inhibitor intraperitoneal injection
  Interventions: Drug: Serplulimab; Drug: Molgramostim; Radiation: Hypofractionated radiotherapy/Sterotactic body radiotherapy

INTERVENTIONS:
Drug: Serplulimab — PD-1 inhibitor (HLX10, serplulimab) 100mg intraperitoneal infusion every two weeks after radiotherapy PD-1 inhibitor (HLX10, serplulimab) 3mg/kg intravenous infusion within one week after radiotherapy every two weeks
  Other Names: HLX10
Drug: Molgramostim — 200ug qd subcutaneous injection for 7 days
  Other Names: rhGM-CSF
Radiation: Hypofractionated radiotherapy/Sterotactic body radiotherapy — 8Gy*3f

SUMMARY:
The effect and safety of intraperitoneal infusion of PD-1 inhibitor is unclear for patients with peritoneal metastasis of advanced malignant tumors and malignant ascites. It is planned to determine the safety and efficacy of intraperitoneal infusion of PD-1 inhibitor combination with PRaG therapy.

DETAILED DESCRIPTION:
Patinets with peritoneal metastasis have limited treatment and poor prognosis. Evidence has shown that there are T lymphocates and macrophages in the ascites microenviroment.We suggested the Intraperitoneal infusion of PD-1 inhibitor might activate T cells and produce anti-tumor effect.The intraperitoneal infusion of PD-1 inhibitorand combined with PRaG(Intravenous injectionof PD-1 inhibitor, Radiotherapy and GM-CSF）might benefit the survival of patients with peritoneal metastasis of advanced malignant tumors with malignant ascites. It is planned to determine the safety in phase I clinical trial. Further through phase II clinical trials, to clarify the effectiveness of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* Pathologically diagnosed malignant tumor abdominal metastasis with malignant ascites (or ascites exfoliative cytology confirmed malignant peritoneal effusion), without brain metastasis or liver metastasis. The patient had newly diagnosed abdominal metastasis with malignant ascites for no more than 1 month.
* Progression on at least one line of prior standard therapy or unsuitability for standard systemic therapy.
* No congestive heart failure, unstable angina pectoris, unstable arrhythmia within the past 6 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-3, and life expectancy 2 months or more.
* No previous severe hematopoietic function, heart, lung, liver, kidney dysfunction and immunodeficiency.
* One week before enrollment, the absolute value of peripheral blood T total lymphocytes ≥ 0.5 times the lower limit of normal, the absolute number of CD8 + T cells ≥ 200/uL, neutrophils ≥ 1.0 × 109/L; AST and ALT ≤ 3.0 times the upper limit of normal; creatinine ≤ 1.5 times the upper limit of normal or creatinine clearance ≥ 50 mL/min, serum albumin ≥ 30 g/L. After treatment, the indicators are allowed to reach the above criteria and last for 2 weeks. Transfusion therapy or granulocyte stimulating factor therapy is not allowed before treatment.
* Patients must have the ability to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with a history of other malignant diseases in the last 2 years, except cured skin cancer and carcinoma in situ.
* Patients with a history of uncontrolled epilepsy, central nervous system diseases or mental disorders, whose clinical severity may hinder the signing of informed consent or affect the patient's compliance with drug treatment as judged by the investigator.
* Clinically significant (ie, active) heart disease, such as symptomatic coronary heart disease, congestive heart failure New York Heart Association (NYHA) Class II or greater, or severe arrhythmia requiring drug intervention, or a history of myocardial infarction within the last 12 months.
* Organ transplantation requiring immunosuppressive therapy.
* Known active infection, or significant hematological, renal, metabolic, gastrointestinal, endocrine function or metabolic disorders, or other serious uncontrolled concomitant diseases as judged by the investigator.
* Hypersensitivity to any component of the study drug.
* History of immunodeficiency, including positive HIV test or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation, or other related diseases requiring long-term oral hormone therapy (greater than 10 mg/d prednisone).
* Patients who are in the period of acute and chronic tuberculosis infection (patients with positive T-spot test and suspicious tuberculosis lesions on chest radiography), are in the period of acute hepatitis infection or have chronic hepatitis B virus copy number higher than the normal range.
* There are contraindications for abdominal paracentesis, including coagulation dysfunction such as severe thrombocytopenia, severe intestinal dilatation and enteroparalysis, and peritoneal adhesion.
* Patients previously treated with immune checkpoint inhibitors and discontinued due to drug-related toxicity.
* Other conditions considered unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT）by CTCAE5.0 | 6 months (phase 1)
  CTCAE is widely accepted throughout the oncology community as the standard classification and severity grading scale for adverse events in cancer therapy clinical trials and other oncology settings
Treatment Related Severe Adverse Effects | 6 months (phase 1)
  Number of participants with treatment-related severe adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
OS | 12 months (phase 2)
  overall survival time

SECONDARY OUTCOMES:
OS | 12 months (phase 1)
  overall survival time
PFS | 12 months (phase 1/2)
  progression-free survival
ascites control rate | 12 months(phase 1/2 )
  ascites control rate

IPD SHARING:
Plan to Share IPD: No